CLINICAL TRIAL: NCT02281903
Title: Is Chest Compressions Using the TrueCPRTM Feedback Device More Effective Than Manual Compressions During Pediatric Resuscitation? A Manikin Study
Brief Title: Pediatric Resuscitation With Feedback CPR Devices
Acronym: PRFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CPR/2014/05
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chest compression of manikins chest (Experimental): Compression of pediatric manikins chest according European Resuscitation Council 2010 guidelines for cardiopulmonary resuscitation.
  Interventions: Device: The TrueCPR feedback device; Device: Standard BLS

INTERVENTIONS:
Device: The TrueCPR feedback device — feedback devices
Device: Standard BLS — Standard basic life support = chest compressions without any feedback device (manual resuscitation)

SUMMARY:
The aim of this study was to compare the TrueCPR feedback device (with metronome) to standard basic life support (BLS) in terms of the quality of single rescuer pediatric resuscitation. Therefore, our hypothesis was that there would be no difference between both CPR methods in terms of chest compression quality parameters.

DETAILED DESCRIPTION:
Cardiac arrest is a leading cause of death worldwide. High-quality chest compressions are of paramount importance for survival and good neurological outcome. Unfortunately, even health professionals have difficulty performing effective CPR. Chest compression (CC) is often too shallow, compression ratio is inadequate, and hands-off time is too long. CPR feedback devices might be an option for rescuers to in order to increase CC efficiency.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* medical profession (paramedics, nurses, physicians) or medical students (nurses, paramedics, physicians)

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Effective compressions compression with correct depth (40-50mm), correct hand position and complete decompressions | 1 month
  effective compressions was defined as compression with correct depth (40-50mm), correct hand position and complete decompressions

SECONDARY OUTCOMES:
effective compressions ratio effective compressions [%] multiplied by flow time [%] | 1 month
  effective compressions ratio was defined as effective compressions [%] multiplied by flow time [%]
Flow time sum of all periods during which chest compressions were performed. | 1 month
  flow time was defined as the sum of all periods during which chest compressions were performed.
absolute hands-off time sum of all periods without chest compressions or ventilation | 1 month
  absolute hands-off time (HOT) was defined as the sum of all periods without chest compressions or ventilation
Compression depth compression in correct depth (40-50mm) measured by the software is connected to the manikin and computer | 1 month
  compression in correct depth (40-50mm) measured by the software is connected to the manikin and computer

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland